CLINICAL TRIAL: NCT04513106
Title: Promoting Advance Care Planning in Persons With Early Stage Dementia and Their Family Caregivers in the Community: a Feasibility Trial
Brief Title: Promoting Advance Care Planning for Persons With Early-stage Dementia in the Community: a Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Chinese University of Hong Kong (Other); The British Council in Hong Kong (Unknown)
Responsible Party: Principal Investigator, Ms Cheryl Yeung Chi Yan, Senior Lecturer, Hong Kong Metropolitan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SIRCP R6303
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Dementia Mild; Mild Cognitive Impairment
Keywords: advance care planning
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participated elderly community centres will be assigned to intervention group or control group at a 1:1 ratio
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group assignment of participants, and the research question.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance care planning programme (Experimental): It is a theory-driven advance care planning programme specifically designed for PWEDs and their family caregivers. The intervention is underpinned by the Bandura's self-efficacy model. Each dyad of participants will receive a 3-session ACP programme, which consists of educational components, guided reflection, and dyadic ACP discussion, guided by ACP facilitators and an ACP booklet. It is composed of 1 group-based sessions and 2 dyadic discussions. One hour for each session, and once weekly. Dyads of participants will be provided with information about the trajectory of dementia, their future healthcare needs and caring options. Their values and care preferences on future care will be elicited in a consistent manner. They will be supported to have an individualized ACP discussion. By the end of the programme, each dyad of participant will be given an ACP booklet documenting the ACP process.
  Interventions: Behavioral: ACP programme "Have a Say"
- Attention control (Placebo Comparator): Dyads of participants in the control group will receive 3-session health talks. One hour for each session, and once weekly. The contents of the health talks are neither dementia-specific nor related to ACP, and cover general health information for elderly, such as drug safety, home safety, exercise and health. This is to differentiate the effect of the intervention from the effect of the extra time and attention given to the participants.
  Interventions: Behavioral: Attention-control health talks

INTERVENTIONS:
Behavioral: ACP programme "Have a Say" — It is a theory-driven advance care planning programme specifically designed for PWEDs or persons with MCI and their family caregivers. The intervention is underpinned by the Bandura's self-efficacy model. Each dyad of participants will receive a 3-session ACP programme, which consists of educational components, guided reflection, and dyadic ACP discussion, guided by ACP facilitators and an ACP booklet. It is composed of 1 group-based sessions and 2 dyadic discussions. One hour for each session, and once weekly. Dyads of participants will be provided with information about the trajectory of dementia, their future healthcare needs and caring options. Their values and care preferences on future care will be elicited in a consistent manner. They will be supported to have an individualized ACP discussion. By the end of the programme, each dyad of participant will be given an ACP booklet documenting the ACP process.
  Arms: Advance care planning programme
Behavioral: Attention-control health talks — Dyads of participants in the control group will receive 3-session health talks. One hour for each session, and once weekly. The contents of the health talks are neither dementia-specific nor related to ACP, and cover general health information for elderly, such as drug safety, home safety, exercise and health. This is to differentiate the effect of the intervention from the effect of the extra time and attention given to the participants
  Arms: Attention control

SUMMARY:
Advance care planning (ACP) has been widely advocated to persons with early stage dementia (PWEDs). This feasibility trial aims to test a theory-based ACP programme "Have a Say" specifically designed for this population, which is underpinned by the Bandura's self-efficacy model. It is the first of its kind in Hong Kong and will be conducted in the community through medical-social collaboration. The aim of this study is to test the feasibility and preliminary effects of the "Have a Say" programme. It is hypothesized that participants in the intervention group will be more engaged in ACP and their dyadic concordance on end-of-life care preference with their family caregivers will be significantly higher than that in the control group.

DETAILED DESCRIPTION:
This study aims to test the feasibility and preliminary effects of an advance care planning (ACP) programme "Have a Say" for persons with early stage dementia (PWEDs) and their family caregivers in the community. A quasi-experimental pretest-posttest study with a control group with repeated blinded outcome assessment will be conducted.

Individuals who have a clinical diagnosis of any form of dementia at the early stage or have a Global Deterioration Score (GDS) 3 or 4 will be eligible to this study. Participated elderly community centres will be assigned to intervention group and control group at 1:1 ratio. Staff members from centres assigned to intervention group will be trained as ACP facilitators and conduct the ACP intervention. Participants in the experimental group will receive a 3-session ACP programme. It includes an educational component, guided reflection and ACP discussion through a series of group-based activity and dyadic discussion delivered by trained ACP facilitator and guided by an ACP booklet. Dyads of participants will be provided with information about the trajectory of dementia, their future healthcare needs and caring options. Their values and care preferences on future care will be elicited in a consistent manner. They will be supported to have an individualized ACP discussion led by ACP facilitators and guided by an ACP booklet. Individuals assigned to the control group will receive attention-control health talks related to ageing. The feasibility of the trial design (in terms of subject recruitment and retention rate) and study instruments (in terms of data completness), and acceptability of intervention procedures (in terms of completion rate and satisfaction score) will be assessed.

As a process evaluation, a group of informants comprised of ACP facilitators and dyads of participants will be conveniently sampled and recruited for an semi-structured individual interview after receiving the intervention. Their experiences of participating in "Have a Say" programme as an ACP facilitator and participants will be explored. Qualitative data will be collected until data saturation. All verbatim will be transcribed and analyzed through qualitative content analysis. The results of this qualitative evaluation will enable us to understand the strengths and weaknesses of this ACP programme during implementation and give us insight about the mechanisms of impact and contextual factors affecting the intervention implementation, sustainability, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* being Chinese,
* being a Cantonese speaker,
* having a formal diagnosis of early stage dementia,
* having a Global Deterioration Scale score 3-4,
* having a designated family caregiver in direct contact.

Exclusion Criteria:

* non-communicable,
* mentally incompetent,
* received an ACP intervention,
* have previously signed an advance directive,
* have other life-limiting chronic illnesses.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in advance care planning engagement | Baseline, immediately after the intervention, 1 month and 3 months follow up
  The behavior change process in ACP behaviours is measured using a 9-item ACP engagement survey. It covers two sub-scales, self-efficacy and readiness, of ACP engagement. Each item is rated on a 5-point likert scale. The higher score means the higher level of engagement for the ACP behaviour.

SECONDARY OUTCOMES:
Change in dyadic concordance of end-of-life care preferences | Baseline, immediately after the intervention, 1 month and 3 months follow up
  The dyadic concordance on end-of-life care preferences is measured by a modified Life Support Preferences Questionnaire (LSPQ). Dyads of participants are invited to answer individually, simultaneously but separately on two hypothetical scenarios, one featured the prospect of developing into advance stage of dementia, and another scenario featured the prospect of developing into an irreversible vegetative stage. PWEDs or persons with MCI are asked to consider themselves in each scenario and indicate their preference for receiving three discrete life-sustaining medical treatments (cardio-pulmonary resuscitation, mechanical ventilation and tube feeding) in each of the two scenarios using a 3 point Likert Scale (want to attempt, refuse or not sure). The dyadic congruence is determined based on whether both of them choose the same option for end-of-life treatments and care goals for the two scenarios. Score ranges from 0-8. A higher score means a higher level of dyadic concordance.
Depression | Baseline, immediately after the intervention, 1 month and 3 months follow up
  The level of depression of PWEDs or persons with MCI is measured by the 19-item Cornell Scale for Depression in Dementia (CSDD). It is to evaluate any adverse outcome posed by the intervention on them. The score ranges from 0-38. A cutoff point of nine or more indicating a depressive disorder, and a higher score means a higher depression level.
Caregivers' stress | Baseline, immediately after the intervention, 1 month and 3 months follow up
  Caregivers' stress is measured by the 12-item Zarit Caregiver Burden Interview. It is to evaluate any adverse outcome posed by the intervention on family caregivers. Score ranges from 0-48. A higher score means a higher level of caregiver burden.

OTHER OUTCOMES:
Subject recruitment rate | Baseline
  The proportion of subjects referred by the centres who were eligible and consented to join the trial
Subject attrition rate | Immediately after the intervention, 1 month and 3 months follow up
  The proportion of subjects consented to the trial and dropout
Completion rate | Immediately after the intervention
  The proportion of subjects completed at least 2 sessions of the intervention out of 3.
Satisfaction score | Immediately after the intervention
  Participants from the intervention group will be asked to complete a 5-item satisfaction questionnaire to provide ratings on the content, timing, and duration of the intervention; the usefulness of the information provided; and the performance of the ACP facilitators. The items are rated on a 5-point Likert scale (5= totally agree; 1= totally disagree), with a higher total score indicating greater satisfaction with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chi Yan Cheryl Yeung, MN, Principal Investigator — Chinese University of Hong Kong
Locations (5):
- Hong Kong (5):
  - Hong Kong Family Welfare Society Kowloon City Centre for Active Ageing, Kowloon
  - Hong Kong Sheng Kung Hui Chuk Yuen Canon Martin District Elderly Community Centre, Kowloon
  - Hong Kong Sheng Kung Hui Lok Man Alice Kwok Integrated Service Centre, Kowloon
  - Yang Memorial Methodist Social Service Choi Hung Community Centre for Senior Citizens, Kowloon
  - Mrs. Wong Tung Yuen District Elderly Community Centre, Yuen Long

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung CC, Ho KH, Chan HY. A dyadic advance care planning intervention for people with early-stage dementia and their family caregivers in a community care setting: a feasibility trial. BMC Geriatr. 2023 Mar 1;23(1):115. doi: 10.1186/s12877-023-03815-3. PMID 36859250